CLINICAL TRIAL: NCT00872872
Title: Nevirapine Plasma Level After Discontinuation of Short-term Antiretroviral Treatment for the Prevention of Mother-to-child Transmission of HIV and Development of Drug Resistant HIV-1 Variants With 1 or 2 Weeks Continuation of Zidovudine/Lamivudine in Women After Delivery
Brief Title: Nevirapine Clearance After Short-term Highly Active Antiretroviral Therapy (HAART) for Prevention of Mother to Child Transmission of HIV (PMTCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Chulalongkorn University (Other); Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-NAT 094
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: NVP Plasma Level; NVP Related Mutation; 3TC Related Mutation
Keywords: NVP; PMTCT; pregnancy; resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZT/3TC 1 week after delivery (Active Comparator): AZT/3TC 1week after delivery
  Interventions: Drug: AZT/3TC 2 weeks after delivery
- AZT/3TC 2 weeks after delivery (Experimental): AZT/3TC 2 weeks after delivery
  Interventions: Drug: AZT/3TC 2 weeks after delivery

INTERVENTIONS:
Drug: AZT/3TC 2 weeks after delivery — AZT/3TC 300/150mg will be given every 12 hours for 1 week after NVP discontinuation in arm 1 and for 2 weeks after NVP discontinuation in arm 2.

SUMMARY:
Three-drug combination of antiretroviral regimens has been used increasingly in HIV-infected pregnant women worldwide, both for the prevention of mother to child transmission of HIV (PMTCT) and for women's own health. Use of these drugs in pregnant women solely for PMTCT means that these drugs will need to be discontinued in the majority of women after delivery.

Certain antiretroviral regimens contain drugs with long half-life (drugs that stay in the body for a longer period of time after discontinuation than other drugs in the same regimen), such as nevirapine (NVP). HIV can easily develop resistance to NVP when NVP is the only drug left in the body (similar to monotherapy). Given two other drugs for up to 1 week after discontinue NVP (to mimic three-drug regimen while waiting for NVP elimination) can help reduce, but not eliminate, the development of resistant virus.

Unfortunately, NVP-containing regimens are the most widely used regimens for pregnant women in developing countries due to its low cost and its availability in fixed-dose combinations. These study will explore how fast NVP is eliminated from women after delivery and to see if given zidovudine/lamivudine (AZT/3TC) for 1 or 2 weeks after NVP discontinuation can help reduce the development of NVP resistant virus.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide 2 separated written informed consents to take part in the Thai Red Cross PMTCT program and in the study
2. Female and aged between 18-45 years
3. Documented HIV-1 infection
4. Pregnant for a maximum of 36 weeks at the first dose of study medication
5. Baseline CD4 cell count >250 cells/mm3
6. Intend to discontinue ART after delivery

Exclusion Criteria:

1. History of significant reaction or allergy to the drugs that may be used in the study
2. Antiretroviral (ARV)-experienced including previous ARV use for the prevention of mother-to-child transmission of HIV
3. Documented NVP- or 3TC-resistant HIV-1 strains
4. Concomitant use of medications that interfere with NVP plasma level
5. Serum aspartate transaminase (AST) or alanine transaminase (ALT) >1.25 times the upper limit of normal
6. Inability to understand the nature and extent of the trial procedures required
7. Pregnant woman, in the opinion of the investigator, should not participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2019-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with detectable NVP plasma level at week 1, 2, 3 and 4 after NVP discontinuation | Week 1, 2, 3 and 4 after NVP discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Thailand